CLINICAL TRIAL: NCT01377415
Title: The Analgesic Effect of Continuous Subacromial Bupivacaine Infusion After Arthroscopic Shoulder Surgery: a Randomized Controlled Trial
Brief Title: Continuous Subacromial Bupivacaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Kari Leino, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: bupi-placebo
Record Dates: First submitted 2011-06-17; First posted 2011-06-21 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Shoulder Arthroscopy
Keywords: arthroscopy; shoulder surgery; subacromial; continuous bupivacaine
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- bupivacaine (Active Comparator): a continuous flow of 5 mg/ml bupivacaine 2 ml/h 48 h
  Interventions: Drug: bupivacaine
- saline (Placebo Comparator): saline 9 mg/ml infusion 2 ml/h 48 h
  Interventions: Drug: bupivacaine

INTERVENTIONS:
Drug: bupivacaine — bupivacaine 5 mg/ml infusion 2 ml/h 48 h
  Other Names: Bicain

SUMMARY:
The investigators wanted to re-evaluate the effects of subacromial bupivacaine infusion after shoulder arthroscopy with standard surgical techniques, including rotator cuff operations. The investigators hypothesized that patients having 5.0 mg/ml bupivacaine infusion at a rate of 2 ml/h subacromially would need less opioids than patients receiving a placebo infusion.

DETAILED DESCRIPTION:
Shoulder surgery has become a routine outpatient procedure. Previously shoulder surgery was associated with intense, occasionally severe postoperative pain and hence considerable use of opioids. Also arthroscopic shoulder surgery, especially rotator cuff procedures, may cause significant pain resulting sometimes in inpatient admission. Subacromial local anaesthetic infusion as a part of a multimodal approach is one commonly used modality to pain relief after shoulder surgery. Nevertheless, it has been criticized recently for its poor benefits and possible adverse effects. On the whole, the scientific evidence of the advantages of local anaesthetic infusions is inconclusive.

ELIGIBILITY:
Inclusion Criteria:

* subacromial impingement disease
* scheduled for an elective arthroscopic surgery

Exclusion Criteria:

* liver disease
* renal impairment
* psychiatric disorder
* alcohol abuse
* obesity (a body mass index of > 35 kg/m2)
* allergies to the drugs used in the study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The consumption of analgesics (oxycodone) | It was recorded on a daily basis during the first three days

SECONDARY OUTCOMES:
The intensity of pain | During the study the pain assessments were recorded 15 min before operation, 15 min, 6, 12 and 18 h after the beginning of the operation and on the first and third postoperative day

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital and University of Turku, Turku, Finland